CLINICAL TRIAL: NCT00387348
Title: Symptom Management Trial in Cancer Survivors
Brief Title: Escitalopram in Treating Depression in Patients With Advanced Lung or Gastrointestinal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB stopped study because placebo arm had more adverse events
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Pirl, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CDR0000505774; MGH-2006-P-000299; K23CA115908 (NIH)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Colorectal Cancer; Depression; Esophageal Cancer; Extrahepatic Bile Duct Cancer; Fatigue; Gallbladder Cancer; Gastric Cancer; Liver Cancer; Lung Cancer; Pancreatic Cancer
Keywords: fatigue; psychosocial effects of cancer and its treatment; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; extensive stage small cell lung cancer; advanced adult primary liver cancer; depression; stage III pancreatic cancer; stage IV pancreatic cancer; stage IV esophageal cancer; stage IV gastric cancer; stage IVA colon cancer; stage IVB colon cancer; stage IVA rectal cancer; stage IVB rectal cancer; unresectable gallbladder cancer; unresectable extrahepatic bile duct cancer
MeSH Terms: conditions — Colorectal Neoplasms; Depression; Esophageal Neoplasms; Bile Duct Neoplasms; Fatigue; Gallbladder Neoplasms; Stomach Neoplasms; Liver Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Rectal Neoplasms | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo-Placebo (Placebo Comparator): Participants in this arm were randomized to receive placebo once daily for the first 4 weeks and placebo once daily for the second 4 weeks
  Interventions: Drug: Placebo
- Placebo-Escitalopram (Other): Participants in this arm were randomized to receive placebo once daily for the first 4 weeks and escitalopram oxalate 10 mg once daily for the second 4 weeks
  Interventions: Drug: escitalopram oxalate; Drug: Placebo
- Escitalopram-Placebo (Other): Participants in this arm were randomzied to receive escitalopram 10 mg once daily for the first 4 weeks and placebo once daily for the second 4 weeks
  Interventions: Drug: escitalopram oxalate; Drug: Placebo

INTERVENTIONS:
Drug: escitalopram oxalate — escitalopram oxalate 10 mg once daily for 4 weeks
  Arms: Escitalopram-Placebo; Placebo-Escitalopram
Drug: Placebo — one placebo pill identical in appearance to the escitalpram pill once daily

SUMMARY:
RATIONALE: Escitalopram may help improve depression and quality of life in patients with advanced lung or gastrointestinal cancer. It is not yet known whether escitalopram is more effective than a placebo in treating depression in patients with advanced lung or gastrointestinal cancer.

PURPOSE: This randomized clinical trial is studying the side effects of escitalopram and to see how well it works compared to a placebo in treating depression in patients with advanced lung or gastrointestinal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of escitalopram oxalate vs placebo in treating major depressive disorder in patients with advanced lung or gastrointestinal cancer.
* Compare the side effect burden of escitalopram oxalate vs placebo in these patients.
* Determine potential moderators of the efficacy of escitalopram oxalate in these patients, including medical, psychological, and social variables.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to stage of disease (stage IIIB with effusions vs stage IV) and current treatment (radiation vs chemotherapy vs novel agent). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral placebo once daily for 4 weeks followed by oral placebo once daily for another 4 weeks
* Arm II: Patients receive oral placebo once daily for 4 weeks followed by escitalopram oxalate 10 mg once daily for 4 weeks.
* Arm III: Patients receive oral escitalopram oxalate 10 mg once daily for 4 weeks followed by oral placebo once daily for 4 weeks.

After 8 weeks, all non-responders are offered open treatment with an antidepressant.

Depression, fatigue, quality of life, anxiety, and somatization are assessed at baseline and then at 4 and 8 weeks.

PROJECTED ACCRUAL: A total of 220 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of any of the following for at least 4 weeks:

  * Stage IIIB (with effusions) or stage IV non-small cell lung cancer
  * Extensive stage small cell lung cancer
  * Stage III or IV pancreatic cancer
  * Stage IV liver cancer
  * Stage III or IV gallbladder cancer
  * Stage III or IV bile duct cancer
  * Stage IV esophageal cancer
  * Stage IV gastric cancer
  * Second line stage IV colorectal cancer
* Meets diagnostic and Statistical Manual of Mental Disorders-4th Edition and Endicott criteria for major depressive disorder
* Duration of depressive symptoms ≥ 4 weeks
* Hamilton Depression D 17 (HAM-D 17) Scale ≥ 14
* No active suicidality requiring immediate care or psychiatric hospitalization

PATIENT CHARACTERISTICS:

* Able to swallow pills
* No active substance abuse disorder (including alcohol abuse within the past 6 months), psychotic disorder or active psychotic symptoms, organic mental disorders, or bipolar disorder
* No clinical or laboratory evidence of hypothyroidism
* No hypercalcemia
* No severe anemia, defined as hemoglobin < 10 g/dL
* No history of multiple adverse drug reactions or allergy to study drugs
* Not pregnant
* No history of head trauma
* No history of epilepsy

PRIOR CONCURRENT THERAPY:

* No other concurrent antidepressant medications or psychostimulants

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William F. Pirl, MD, Study Chair — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the ambulatory thoracic and GI cancer clinics at MGH. Recruitment was open from 11/1/06 until 4/1/11.
Pre-assignment Details: After enrollment, participants completed an assessment for major depressive disorder. 90 participants consented for study evaluation. In order to be randomized to a group, participants had to meet criteria for major depressive disorder. Of the 90 evaluated on study, only 24 were randomized.
Groups:
- Placebo-Placebo: Participants in this arm were randomized to receive placebo once daily by mouth for the first 4 weeks and placebo once daily by mouth for the second 4 weeks.
- Placebo-Escitalopram: Participants in this arm were randomized to receive placebo once daily by mouth for the first 4 weeks and escitalopram 10 mg once daily by mouth for the second 4 weeks
- Escitalopram-Placebo: Participants in this arm were randomzied to receive escitalopram 10 mg once daily by mouth for the first 4 weeks and placebo once daily by mouth for the second 4 weeks
Period: Overall Study
Arm/Group | Placebo-Placebo | Placebo-Escitalopram | Escitalopram-Placebo
Started | 8 | 5 | 11
Completed | 5 | 2 | 7
Not Completed | 3 | 3 | 4
Not completed — Death | 1 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo-Placebo: Participants in this arm were randomized to receive placebo for the first 4 weeks and placebo for the second 4 weeks
- Placebo-Escitalopram: Participants in this arm were randomized to receive placebo for the first 4 weeks and escitalopram for the second 4 weeks
- Escitalopram-Placebo: Participants in this arm were randomzied to receive escitalopram for the first 4 weeks and placebo for the second 4 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo-Placebo | Placebo-Escitalopram | Escitalopram-Placebo | Total
Number analyzed (Participants) | 8 | 5 | 11 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 8 | 19
  >=65 years | 1 | 1 | 3 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 56.63 (10.51) | 59.40 (10.84) | 58.36 (9.41) | 58.00 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7 | 14
  Male | 4 | 2 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Depression Response Rate of Escitalopram Oxalate 10 mg Once Daily Compared to Placebo Once Daily for Major Depressive Disorder
Description: Response rate was defined as a 50% reduction in the Hamilton Depression Rating Scale (HAM-D) scores over 4 weeks. The HAM-D can have total scores that range from 0 to 50, with higher scores indicating greater depression. Scores over 14 are considered to be in the depressed range.
Time Frame: 4 weeks
Population: The efficacy analysis was intent to treat and all randomized participants were analyzed
Measure: Number; unit: number of participants with response
Groups:
- Placebo-Placebo: Participants in this arm were randomized to receive placebo once daily by mouth for the first 4 weeks and placebo oncedaily by mouth for the second 4 weeks
- Escitalopram-Placebo: Participants in this arm were randomzied to receive escitalopram f10 mg once daily by mouth or the first 4 weeks and placebo once daily by mouth for the second 4 weeks
Arm/Group | Placebo-Placebo | Placebo-Escitalopram | Escitalopram-Placebo
Number analyzed (Participants) | 8 | 5 | 11
number of participants with response | 3 (0.52) | 1 (0.47) | 6 (0.52)

2. Secondary Outcome: Side Effect Burden
Description: Side efect burden was defined as the total score of the UKU Side Effects Rating Scale. This scale contains 48 items corresponding to side effects which are rated from 0-3, with 0 meaning not present and 1-3 rating the severity of the side effect. Higher scores represented greater side effect burden. The scale range is 0 to 144.
Time Frame: 4 weeks
Population: Participants who completed the 4 week assessment were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo-Placebo | Placebo-Escitalopram | Escitalopram-Placebo
Number analyzed (Participants) | 6 | 2 | 9
units on a scale | 3.00 (2.10) | 2.50 (0.71) | 3.44 (1.88)

3. Primary Outcome: Change in Hamilton Depression Rating Scale (HAM-D) Scores
Description: The change in HAM-D scores was calculated by subtracting the score at 4 weeks from the score at baseline. The HAM-D can have total scores that range from 0 to 50, with higher scores indicating greater depression. Scores over 14 are considered to be in the depressed range.
Time Frame: 4 weeks
Population: Participants who had at least 1 follow up HAM-D assessment were included. Two participants died, one without a follow up assessment and one with a HAM-D at 2 weeks. For the participant who had the HAM-D at 2 weeks and then died, the last endpoint was carried forward.
Measure: Mean (Standard Deviation); unit: Change in HAM-D scores
Arm/Group | Placebo-Placebo | Placebo-Escitalopram | Escitalopram-Placebo
Number analyzed (Participants) | 7 | 5 | 11
Change in HAM-D scores | 6.23 (8.37) | 10.60 (5.18) | 6.45 (5.18)

ADVERSE EVENTS:
Arm/Group | Placebo-Placebo | Placebo-Escitalopram | Escitalopram-Placebo
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/5 | 0/11
Other Adverse Events (participants affected / at risk) | 1/8 | 0/5 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-Placebo (N=8) | Placebo-Escitalopram (N=5) | Escitalopram-Placebo (N=11)
death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-Placebo (N=8) | Placebo-Escitalopram (N=5) | Escitalopram-Placebo (N=11)
HAM-D score increased by at least 25% (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
After an interim analaysis, the DSMB decided to terminate the trial early because of the rate of adverse events (HAM-D scores increasing by at least 25%) and deaths were higher in participants receiving placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No